CLINICAL TRIAL: NCT04551235
Title: Establishing Automatic Method of Counting and Classify Bone Marrow and Peripheral Blood Cells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Tai-Chen Cell Therapy Center, Biomdcare Corporation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202007086RIPB
Record Dates: First submitted 2020-08-27; First posted 2020-09-16 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Hematologic Diseases; Artificial Intelligence; Acute Leukemia
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: there are not any interventions in this study — there are not any interventions in this study

SUMMARY:
Counting and classification of blood cells in a bone marrow smear and peripheral blood smear are essential to clinical hematology. To this date, this procedure has been carried out in a manual manner in the great majority of clinical settings. There is often inconsistency in the counting result between different operators largely due to its manual nature. There has not been an effective and standard method for blood smear preparation and automatic counting and classification. The recent advent of deep neural network for medical image processing introduced new opportunities for an effective solution of this long-standing problem. Numerous results have been published on the effectiveness of convolutional neural network in clinical image recognition task.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have suspected or confirmed hematological diseases and receive bone
* marrow or peripheral blood cell morphological examination in National Taiwan University Cancer Center
* Patients who are aged more than 20 y/o

Exclusion Criteria:

•Patients who are not willing to sign informed consents

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have suspected or confirmed hematological diseases and receive bone marrow or peripheral blood cell morphological examination in National Taiwan University Cancer Center
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the accuracy of cell counting and classifying between automatic method and manual method through digital microscopic photos of bone marrow smear and peripheral blood smear using deep convolutional neural networks | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Tai-Chen Cell Therapy Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided